CLINICAL TRIAL: NCT06293404
Title: The Effect of Spinal Column Flexion on Unilaterality of Spinal Anesthesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: column flexion; AnkaraCHBilkent (Other: AnkaraCHBilkent)
Record Dates: First submitted 2024-01-31; First posted 2024-03-05 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Hip Fractures; Spinal Anesthesia
Keywords: position effect; hip fracture; spinal anesthesia
MeSH Terms: conditions — Hip Fractures | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group F (Active Comparator): the lateral decubitus position, Group F will keep the spinal cord flexed for 10 minutes,
  Interventions: Drug: Bupivacain
- Group N (Other): the lateral decubitus position, Group N will keep the natural position of the spinal cord in lateral decubitus for 10 minutes,
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Bupivacain — 7.5 mg Bupivacaine hydrochloride (0.5% heavy Marcaine) will be used on spinal anesthesia. (each group)

SUMMARY:
The effect of two different positions on spinal anesthesia in hip fracture surgery

DETAILED DESCRIPTION:
One of the more common reasons for hospitalization in affluent nations is femoral fractures. Postpartum mortality and morbidity rates for femur fractures are significant. Mortality rates range from 5% to 8% at the time of initial admission and from 14% to 36% throughout the first year. Age-related mortality rates are rising. Surgery is necessary for femur fractures, and spinal anesthesia is frequently the recommended anaesthetic approach.

After spinal anesthesia, hypotension is frequently seen as a result of sympathetic block and a reduction in systemic vascular resistance. The frequency of hypotension rises as the level of spinal anesthetic block increases, especially in older people. It has been demonstrated that hypotension is connected with an increased mortality rate.

Preoperative fluid administration to reduce hypotension loading, lateral decubitus anesthesia posture, and spinal anesthetic dose reduction techniques have all been used.

There are several methods to enhance the quality of the block in spinal anesthesia, including local changes to the anesthetic's baricity, volume, infusion rate, and lateral decubitus position. There are numerous variables, including residency time and spinal needle type. The influence of alterations in the spinal cord inside the vertebral column on body position in the literature was examined using lumbar MR imaging. Based on these research, it was intended to study the role that alterations in spinal anesthesia played in the applications of spinal anesthesia. spinal column Hemiblock is thought to result in more stable hemodynamics during anesthesia. Studies can be found. The goal of this study is to administer semispinal anesthesia while doing spinal anesthesia. To ensure that the underlying spinal cord is impacted by the local anesthetic and to monitor the impact on unilateral block development and hemodynamic parameters, the colon is flexed and squeezed to the surgery side and anterior area of the spinal cord.

The study will take unilateral femoral fracture surgery into account. Both groups will be given spinal anesthesia in the study's lateral

First, Group F will keep the spinal cord flexed for 10 minutes while Group N will preserve the spinal cord's normal position in lateral decubitus. The quality of the ensuing block will be compared between the two groups. When spinal anesthetic is being used, patients may feel excruciating pain while in the prescribed position.

To lessen positional pain and the impact of hemodynamic deterioration brought on by pain during spinal anesthesia, pericapsular nerve group (PENG) block will be used.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2-3
* Hip fracture
* 18-85 Age
* BMI: 18-40

Exclusion Criteria:

* ASA score of 4 and above
* Left ventricular ejection fraction below 40%
* Severe aortic valve stenosis
* Obesity (BMI >40)
* Presence of cardiac arrhythmia
* Having peripheral vascular disease
* Failure of spinal block
* Bleeding diathesis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic change | Within 3 minutes after anesthesia
  Heart rate
Hemodynamic change | Within 5 minutes after anesthesia
  Heart rate
Hemodynamic change | Within 10 minutes after anesthesia
  Heart rate
Hemodynamic change blockade to the dependent lower limb in flexed and extended spine position. | 15 minutes
  Heart rate
Hemodynamic change blockade to the dependent lower limb in flexed and extended spine position. | 20 minutes after anesthesia
  Heart rate
Hemodynamic change blockade to the dependent lower limb in flexed and extended spine position. | 30 minutes after anesthesia
  Heart rate

SECONDARY OUTCOMES:
To compare the efficacy, duration of motor block until return to normal function in the non-operated leg after the start of injection, of bupivacaine 7.5 mg/ml when used for spinal anaesthesia in patients undergoing unilateral lower | 10 minutes after anesthesia
  bromage score

OTHER OUTCOMES:
To compare the efficacy of bupivacaine 7.5 mg/ml in the duration of sensory block at dermatome T10 level | Within 1 minutes after anesthesia
  sensory block time

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sahap, Study Director — Ankara City Hospital Bilkent

IPD SHARING:
Plan to Share IPD: No
only results